CLINICAL TRIAL: NCT00889044
Title: Chewing Clopidogrel in Addition to Regular Oral Clopidogrel Treatment to Improve Platelets Aggregation in Patient With NON ST ELEVATION MI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Shlomi Matetzky, Sheba Medical Center
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHEBA-08 -5397-SM-CTIL
Record Dates: First submitted 2009-04-26; First posted 2009-04-28 (Estimated); Last update posted 2009-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Platlet Aggregation; Major Bleeding Outcomes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- clopidogrel by chewing (Experimental)
  Interventions: Drug: clopidogrel by chewing
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: clopidogrel by chewing — 600 mg clopidogrel by chewing
  Arms: clopidogrel by chewing
Drug: Placebo — Placebo p.o
  Arms: Placebo

SUMMARY:
Since the absorption of clopidogrel through the gastrointestinal tract is limited, we want to examine whether adding clopidogrel by chewing will overcome the limited gastrointestinal absorption, and hence will improve the prevention of platelet aggregation.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female older than 18 years old with non-ST myocardial infarction

Exclusion Criteria:

* Current treatment with anticoagulation medication, any type of cerebro vascular event in the past, active bleeding, active peptic ulcer disease, pregnant women, any inability to sign an informed consent of participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Platelet aggregation and bleeding events | 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Sheba Medical Center, Cardiac Institute, Tel Litwinsky, Tel Hashomer
  - Sheba_medical_center, Ramat Gan

REFERENCES:
- [Background] Gurbel PA, Bliden KP, Hiatt BL, O'Connor CM. Clopidogrel for coronary stenting: response variability, drug resistance, and the effect of pretreatment platelet reactivity. Circulation. 2003 Jun 17;107(23):2908-13. doi: 10.1161/01.CIR.0000072771.11429.83. Epub 2003 Jun 9. PMID 12796140
- [Background] Matetzky S, Shenkman B, Guetta V, Shechter M, Beinart R, Goldenberg I, Novikov I, Pres H, Savion N, Varon D, Hod H. Clopidogrel resistance is associated with increased risk of recurrent atherothrombotic events in patients with acute myocardial infarction. Circulation. 2004 Jun 29;109(25):3171-5. doi: 10.1161/01.CIR.0000130846.46168.03. Epub 2004 Jun 7. PMID 15184279